CLINICAL TRIAL: NCT04831736
Title: Randomized, Single-blind, Placebo-controlled Study on the Effect of Postoperative Administration of Single Dose Ketamine After Mastectomy on Pain
Brief Title: Effect of Postoperative Single Dose of Ketamine on Pain After Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-00072
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
Keywords: Mastectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Ketamine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine at a dose of 0.6 mg/kg will be administered intravenously (IV) while the participant is recovering in the PACU. The study drug will be administered over at least 30 minutes at one time point and will be administered after subject has been deemed to be stable (hemodynamically stable, awake) by the study team on POD 0.
  Arms: Treatment
Drug: Placebo — Matching equal dose of saline placebo will be administered intravenously while the participant is recovering in the PACU.
  Arms: Control

SUMMARY:
This is a randomized, single blinded, placebo-controlled trial to study the effectiveness of a subanesthetic dose (0.6mg/kg) of ketamine versus placebo (saline) on postoperative pain on adult women undergoing mastectomy.

The objective of the study is to examine the effect of a subanesthetic dose (0.6mg/kg) of ketamine vs. saline control on postoperative pain in subjects who have undergone mastectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women, aged 18 to 80 years old, who will undergo mastectomy.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Will be scheduled for elective breast surgery for oncologic indication as follows: mastectomy +/- lymph node dissection, prophylactic mastectomy, unilateral or bilateral, with immediate reconstruction
4. No distant metastases.
5. Subject is American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
6. Subject is medically stable.

Exclusion Criteria:

1. Cognitive impairment (by history) or clinical signs of altered mental status such as confusion, amnesia, disorientation, fluctuating levels of alertness, etc. that may interference with adherence to study procedures and/or participant safety.
2. Past ketamine or phencyclidine misuse or abuse.
3. Schizophrenia or history of psychosis.
4. Known sensitivity or allergy to ketamine.
5. Liver or renal insufficiency.
6. History of uncontrolled hypertension, chest pain, cardiac arrythmia, stroke, head trauma, intracranial mass or hemorrhage or pressure, glaucoma, acute globe injury, uncontrolled thyroid disease, porphyria, or any other contraindication to ketamine. Use of lamotrigine, alfentanil, physostigmine, and 4-aminopyridine are contraindicated
7. Pregnancy or nursing women
8. BMI>35.
9. Currently participating in another pain interventional trial.
10. Unwillingness to give informed consent.
11. Non-English speaking patients as QoR-15 and BCPQ have not been validated in all other languages

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Doan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to lisa.doan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 15 | 16
Completed | 15 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 48.9 [25 to 62] | 46.5 [32 to 73] | 47.3 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory-short Form (BPI) Pain Severity Subscale Score
Description: BPI Pain Severity Subscale consists of 4 questions (asking to rate pain). Each question is answered on a scale 0 (no pain) to 10 (pain as bad as you can imagine). The total range of score is 0-40; the higher the score, the worse the pain.
Time Frame: 24 Hours Post-Op (Day 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 16.7 (6.97) | 18.1 (8.44)

2. Primary Outcome: Brief Pain Inventory-short Form (BPI) Pain Severity Subscale Score
Description: as for outcome 1
Time Frame: 48 Hours Post-Op (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 16 (5.32) | 15.7 (9.36)

3. Secondary Outcome: Brief Pain Inventory-short Form (BPI) Pain Severity Subscale Score
Description: BPI Pain Severity Subscale is a 4-item questionnaire asking participants to rate pain. Each question is answered on a scale 0 (no pain) to 10 (pain as bad as you can imagine). The total range of score is 0-40; the higher the score, the worse the pain.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 3.5 (6.45) | 2.2 (5.37)

4. Secondary Outcome: Brief Pain Inventory-short Form (BPI) Pain Severity Subscale Score
Description: as for outcome 3
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 11.5 (6.17) | 15 (8.68)

5. Secondary Outcome: Brief Pain Inventory-short Form (BPI) Pain Interference Subscale Score
Description: BPI Pain Interference Subscale is a 7-item questionnaire asking participants to describe how pain has interfered during activities. Each question is answered on a scale 0 (does not interfere) to 10 (completely interferes). The total range of score is 0-70; the higher the score, the worse the interference.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 4 | 3
score on a scale | 35 (18.29) | 35 (30.35)

6. Secondary Outcome: Brief Pain Inventory-short Form (BPI) Pain Interference Subscale Score
Description: as for outcome 5
Time Frame: Day 1 Post-Op (Day 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 24.7 (17.1) | 28.1 (14.9)

7. Secondary Outcome: Brief Pain Inventory-short Form (BPI) Pain Interference Subscale Score
Description: as for outcome 5
Time Frame: Day 2 Post-Op (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 33.5 (12.5) | 32.1 (15.5)

8. Secondary Outcome: Brief Pain Inventory-short Form (BPI) Pain Interference Subscale Score
Description: as for outcome 5
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 33.9 (18.3) | 32.9 (15.1)

9. Secondary Outcome: Total Dosage of Opioid Use
Description: Use and dosage will be assessed through medical records and subject reports.
Time Frame: Day of Surgery (Day 1)
Measure: Mean (Standard Deviation); unit: oral morphine equivalent (mg)
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
oral morphine equivalent (mg) | 6 (7.06) | 5 (6.61)

10. Secondary Outcome: Total Dosage of Opioid Use
Description: Use and dosage will be assessed through medical records and subject reports.
Time Frame: Day 1 Post-Op (Day 2)
Measure: Mean (Standard Deviation); unit: oral morphine equivalent (mg)
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
oral morphine equivalent (mg) | 21.5 (17.9) | 37.2 (61.4)

11. Secondary Outcome: Total Dosage of Opioid Use
Description: Use and dosage will be assess through medical records and subject reports.
Time Frame: Day 2 Post-Op (Day 3)
Measure: Mean (Standard Deviation); unit: oral morphine equivalent (mg)
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
oral morphine equivalent (mg) | 21.2 (31.1) | 18.5 (21.2)

12. Secondary Outcome: Total Dosage of Opioid Use
Description: Use and dosage will be assess through medical records and subject reports.
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: oral morphine equivalent (mg)
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
oral morphine equivalent (mg) | 0.833 (2.25) | 7 (2.25)

13. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (Short Form 7b) Daily Score
Description: The PROMIS Fatigue Short Form consists of 7 questions evaluating the frequency of fatigue. Each question is answered with a score from 1 (never) to 5 (always). The raw score is the sum of each item and ranges from 7-35. Raw scores are converted to T-scores ranging from 31 to 81.4, with a standard deviation of 10. Higher T-scores indicate higher frequency of fatigue.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
T-score | 46.7 (12.5) | 44.5 (9.51)

14. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (Short Form 7b) Daily Score
Description: as for outcome 13
Time Frame: Day 1 Post-Op (Day 2)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
T-score | 52.3 (13.1) | 53.6 (10.5)

15. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (Short Form 7b) Daily Score
Description: as for outcome 13
Time Frame: Day 2 Post-Op (Day 3)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
T-score | 56.6 (7.07) | 54 (7.71)

16. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (Short Form 7b) Daily Score
Description: as for outcome 13
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
T-score | 49.1 (10.6) | 50.4 (10.8)

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (Short Form 6A) Score
Description: The PROMIS Sleep Disturbance Short Form consists of 6 items assessing sleep disturbance. Each question is answered with a score of 1-5 (varies). The raw score is the sum of each item and ranges from 6-30. The raw score is converted to a T-score ranging from 31.7 to 76.1, with a standard deviation of 10. Higher T-scores indicate greater sleep disturbance.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
T-score | 53.6 (5.39) | 49.2 (10.1)

18. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (Short Form 6A) Score
Description: as for outcome 17
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
T-score | 51.7 (9.19) | 50.7 (9.2)

19. Secondary Outcome: Generalized Anxiety Disorder (GAD-2) Score
Description: GAD-2 consists of 2 items and measures how often one has been bothered by anxiety-related problems. Each is answered with a score of 0 (not at all) to 3 (nearly every day). The total range of score is 0-6; the higher the score, the more frequent one is bothered by anxiety.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 2.47 (1.77) | 1.87 (2.07)

20. Secondary Outcome: Generalized Anxiety Disorder (GAD-2) Score
Description: as for outcome 19
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 2.13 (1.73) | 1.13 (1.51)

21. Secondary Outcome: Breast Cancer Pain Questionnaire (BCPQ) - Pain Score
Description: If the patient reports pain in the area of the breast, armpit, side of the body, or arm on the side of operation, the patient will be asked to report level of pain (0 is no pain and 10 is the worst pain imaginable). For each location, the total score is 0-10; the higher the score, the worse the pain. The total score is the sum of responses from each location.
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 3.53 (2.56) | 4.6 (2.72)

22. Secondary Outcome: Quality of Recovery (QoR-15) Survey Score
Description: Part A of QoR-15 consists of 10 conditions. Based on how the patient has been feeling in the last 24 hours, they will respond to each condition using an 11-point Likert scale ranging from 0 to 10, where 0 is none of the time [poor] and 10 is all of the time [excellent]). The total range of score for Part A is 0-100; the higher the score, the better the participant has been feeling.
  Part B consists of 5 symptoms. The patient will indicate whether they have experienced each symptom over the last 24 hours using an 11-point Likert scale ranging from 10 to 0, where 10 is none of the time [excellent] and 0 is all of the time [poor]). The total range of score for Part B is 0-50; the higher the score, the better the participant has been feeling.
  The total score is the sum of of scores from Parts A and B. Total scores range from 0-150; the higher the score, the better the participant has been feeling.
Time Frame: Day 2 Post-Op (Day 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 75.1 (12) | 74.6 (13.2)

23. Secondary Outcome: Quality of Recovery (QoR-15) Survey Score
Description: Part A of QoR-15 consists of 10 conditions. Based on how the patient has been feeling in the last 24 hours, they will respond to each condition using an 11-point Likert scale ranging from 0 to 10, where 0 is none of the time [poor] and 10 is all of the time [excellent]). The total range of score for Part A is 0-100; the higher the score, the better the participant has been feeling.
  Part B consists of 5 symptoms. The patient will indicate whether they have experienced each symptom over the last 24 hours using an 11-point Likert scale ranging from 10 to 0, where 10 is none of the time [excellent] and 0 is all of the time [poor]). The total range of score for Part B is 0-50; the higher the score, the better the participant has been feeling.
  The total score is the sum of of scores from Parts A and B. Scores range from 0-150; the higher the score, the better the participant has been feeling.
Time Frame: Day 7 Post-Op (Day 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
score on a scale | 81.6 (18.4) | 80.4 (11.5)

24. Secondary Outcome: Number of Participants Who Experience Side Effects
Description: Side effects are calculated using a 7-item psycho-behavioral questionnaire. Participants indicate whether they have experienced any of the listed side effects of ketamine. The side effects listed on the questionnaire are not considered to be Adverse Events or Serious Adverse Events.
Time Frame: Day of Surgery (Day 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
Participants | 7 | 7

25. Secondary Outcome: Number of Participants Who Experience Side Effects
Description: Side effects are calculated using a 7-item psycho-behavioral questionnaire. Participants indicate whether they have experienced any of the listed side effects. The side effects listed on the questionnaire are not considered to be Adverse Events or Serious Adverse Events.
Time Frame: Day 1 Post-Op (Day 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 7 Days
Description: Participants self-reported adverse events. Side effects reported using the 7-item psycho-behavioral questionnaire (see Outcome Measures #24 and #25) were not considered to be Adverse Events or Serious Adverse Events.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT04831736/Prot_SAP_000.pdf